CLINICAL TRIAL: NCT07036081
Title: A Single Arm Intervention Study to Assess the Acceptability, Tolerance and Ease of Use of Wilbo's Blends+ (Commercial Enteral Feed Based on Real Food) When Used as Part of a Dietitian Prescribed Enteral Feeding Plan
Acronym: Wilbo's Blends
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Manchester (Other); Wilbo's Blends (Unknown); Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24CS011; IUK10068044 (Other Grant/Funding Number: Innovate UK)
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: Enteral Nutrition (Food for Special Medical Purposes); Enteral Feeds; Enteral Tube Nutrition; Gastrostomy Tube
Keywords: Enteral Tube Feeding; Gastrostomy Tube; Enteral Nutrition; Enteral Formula; Enteral Feeds

STUDY DESIGN:
Intervention Model Description: Participant's selection will be made by purposive sampling following the eligibility criteria and clinician/dietitians' recommendation. Participants will be invited into clinic or via the Home Enteral Feeding service home visits (in accordance with local practice) to consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- • Children and young people (age 3-15) who are assessed by a Doctor or Dietitian as requiring entera (Experimental): A new feeding plan will be developed by the study dietitians. Participants will be transitioned from their current enteral feeding plan to incorporate Wilbo's Blends+. In this new plan Wilbo's Blends+ can provide up to 100% but not lower than 30% of their total daily calorie requirements depending on participant's individual clinical needs, as assessed by the study dietitian.
  Interventions: Dietary Supplement: Wilbo's Blends+

INTERVENTIONS:
Dietary Supplement: Wilbo's Blends+ — A new feeding plan will be developed by the study dietitians. Participants will be transitioned from their current enteral feeding plan to incorporate Wilbo's Blends+. In this new plan Wilbo's Blends+ can provide up to 100% but not lower than 30% of their total daily calorie requirements depending on participant's individual clinical needs, as assessed by the study dietitian.
  All participants will be on at least 30% Wilbo's Blends+ for at least 7 days.
  If required clinically there is the option to transition participants onto Wilbo's Blends+ over 1-6 days, for children who are deemed particularly sensitive to change in their feeding plan.
  Participants or their families/carers will complete an electronic workbook consisting of:
  * GI tolerance records for 7 days whilst receiving Wilbo's Blends+
  * Compliance records for 7 days whilst receiving Wilbo's Blends+
  * Ease of use and palatability questionnaire at the end of the study intervention (after last administration of Wilbo's Blends+

SUMMARY:
The goal of this observational study is to learn if tube-fed children and young people (age 3-15 years) find Wilbo's Blends+ (a new nutritionally complete enteral formula containing real food ingredients) acceptable, tolerable and easy to use. The main question it aims to answer is:

Is Wilbo's Blends+ acceptable when included in the feeding plan of tube-fed children and young people (age 3-15 years)

Participants will:

Take Wilbo's Blend+ for a 7 day period as part of their feeding plan Complete questionnaires about their gastrointestinal symptoms

DETAILED DESCRIPTION:
THEORETICAL FRAMEWORK The study design follows the UK Advisory Committee on Borderline Substances (ACBS) criteria to support submission for prescription usage in the National Health Service (NHS).

RESEARCH QUESTION / AIM(S) Is a commercially prepared nutritionally complete enteral formula made with real food ingredients accepted, tolerated and complied with instead of a patient's usual enteral formula?

Objectives

Primary:

To test the acceptability of Wilbo's Blends+ with regards to GI tolerance and compliance, following UK ACBS criteria to support submission for prescription usage in the NHS.

Secondary:

* To test ease of use of the Wilbo's Blends+ product.
* To test where possible palatability of the Wilbo's Blends+ product.
* To record the food, feed, and fluid intake while taking Wilbo's Blends+ as part of a Dietitian prescribed enteral feeding plan.
* To collect data on Health Care Team perceptions of the child's tolerance to Wilbo's Blends+.

STUDY DESIGN AND METHODS OF DATA/SAMPLE COLLECTION AND DATA/SAMPLE ANALYSIS

Study Design The study design follows the UK Advisory Committee on Borderline Substances (ACBS) criteria to support submission for prescription usage in the NHS.

This will be a prospective, open-label single arm interventional study that will use participant/parent/carer-reported questionnaires and records alongside Case Report Forms (CRFs) completed by the clinical team for data collection.

Methods of Data Collection The CI will assign participants with a study ID at the stage of consent. There will be an MS Excel spreadsheet which holds the pseudonymised ID and the individuals' names in case a participant needs to be re-identified for any reason. This is called the pseudonymisation key. This will be kept safe in a password protected shared area which is separate to the rest of the study documentation. The spreadsheet should have audit tracking enabled.

The demographic data should be stored only with the study ID on a password protected MSExcel spreadsheet with audit tracking enabled. This will be collected and inputted by the study team from the participant's medical records. This will be kept safe in a password protected shared area which is accessible only to the study team.

The CRF is paper, and will be linked to the participant via their study ID. All data collected at the baseline and follow-up visit and perceptions of the participant's clinical team prior to and following use of Wilbo's Blends+ will be captured using the CRFs. The managing dietitian/member of the clinical team (who knows the patient) will complete the baseline questionnaire using reports from the participant/parent/carer and medical notes. The data from the paper CRF will be transcribed onto a MS Excel spreadsheet during the study. This will be kept safe in a password protected shared area which is accessible only to the study team. The spreadsheet should have audit tracking enabled.

All participant questionnaires (the workbook) will be in electronic format (Jisc). Paper versions can be made available on request and will be returned to the study team at the end of the study using the provided stamped addressed envelopes or at the follow-up visit. Paper versions will be transcribed into a MS Excel spreadsheet by the site study team. The original copy must be maintained at site and kept in a locked cabinet in a secure room which is accessible only to the study team (as this is source data). Any study workbooks completed on Jisc will be exported onto a MS Excel spreadsheet throughout the study and saved in a secure/restricted access area of the shared drive. The spreadsheet should have audit tracking enabled. The study team at MFT will need to scan and email paper CRFs, study workbooks, and MS Excel spreadsheet to the Trial Manager using secure NHS encrypted email. This is so the Trial Manager can complete a quality control check on the transcription. The Trial Manager will complete NUH checks in person where possible.

Data will be kept for the duration of the study, plus the study write up period, which totals 2 years. All study data will then be anonymised and archived. After 5 years, it will be destroyed according to R&I SOPs.

STUDY SETTING This is a multicentre study with two recruiting sites - Nottingham University Hospitals NHS Trust and Manchester Foundation Trust.

Sampling technique Participant's selection will be made by purposive sampling following the eligibility criteria and clinician/dietitians' recommendation. Participants will be invited into clinic or via the Home Enteral Feeding service home visits (in accordance with local practice) to consent.

Recruitment Participants will be identified by existing members of the participant's clinical care team as meeting the eligibility criteria during the participant's routine NHS care and via pre-screening patient lists. The clinical team will ask whether family/carers/participants are happy to be contacted and once this has been agreed they will be approached to take part by the Principal Investigator or dietitian (all those approaching will have Good Clinical Practice training). There is no plan to recruit through publicity i.e. posters or patient identification centres.

Parent/carers will be provided with an information sheet and consent form. Participants will be given an age-appropriate Participant Information Sheet (PIS) and assent form and invited back to clinic/a home visit organised > 24 hours after receipt to be screened and consented if eligibility criteria are met.

Sample identification Participants who meet the eligibility criteria will be identified by a member of their existing clinical care team through routine outpatient follow up or inpatient monitoring. They and their parents/carers will be provided with the relevant PISs.

Consent Potential participants' parents/carers will be contacted by phone no less than 24 hours after receiving the PIS, and if they wish to consent, a baseline visit will be arranged. There will be discussion between the potential participant and his/her legally acceptable representatives (parent/carer) and the Principal Investigator or nominated study representative as detailed on the study delegation log about the nature and objectives of the study and possible risks. Parent/carers will provide consent and participants will provide assent. A verbal assent form can be used for some participants who have disabilities which render them unable to complete a physical assent form, and a verbal consent form is available for parent/carers. Upon completion of consent and assent, further eligibility checks and baseline assessments will be conducted and a dietetic plan incorporating Wilbo's Blends+ produced for the participant. All consent and assent will be taken on paper copies.

The Wilbo's Blends+ product will be distributed directly to the Participant's home address by Wilbo's Blends. Participants will receive the packages of Wilbo's Blends+ product with instructions, recommendations, and contact information. If they do not wish for it to be delivered to their home address, it can be arranged that they collect this from the hospital.

Study Assessments A new feeding plan will be developed by the study dietitians. Participants will be transitioned from their current enteral feeding plan to incorporate Wilbo's Blends+. In this new plan Wilbo's Blends+ can provide up to 100% but not lower than 30% of their total daily calorie requirements depending on participant's individual clinical needs, as assessed by the study dietitian.

All participants will be on at least 30% Wilbo's Blends+ for at least 7 days.

If required clinically there is the option to transition participants onto Wilbo's Blends+ over 1-6 days, for children who are deemed particularly sensitive to change in their feeding plan.

Participants or their families/carers will complete an electronic workbook consisting of:

* GI tolerance records for 7 days whilst receiving Wilbo's Blends+
* Compliance records for 7 days whilst receiving Wilbo's Blends+
* Ease of use and palatability questionnaire at the end of the study intervention (after last administration of Wilbo's Blends+).

Day 1 of receiving Wilbo's Blends+ can take place up to 14 days after the screening and consent visit as long as there have not been any changes in baseline symptoms or hospitalisations and the end of study questionnaire and visit can be up to up to 6 days after finishing Wilbo's Blends+.

After the 7 days of Wilbo's Blends+ participants return to their pre-study feeding plan. There is no provision to supply study product after the 7-day period, however participants will be offered a 20% discount code (cost value) on the Wilbo's Blends existing product range until an ACBS decision has been made.

Participants with missing data will be followed up for completion. If the data is not completed/returned, then that participant will be replaced.

Long term follow-up assessments This is an acceptability study over a short intervention period. Following the end of study visit (at day 14-18 in clinic or over telephone/video), no long-term follow up is required.

Withdrawal Criteria Participants will be withdrawn from the study if they are admitted to hospital or unwell for any reason relating to their underlying medical condition during the 7 days of receiving Wilbo's Blends+.

Parents/carers are able to withdraw their child from the study at any point. If a participant is withdrawn from the study the reasons for withdrawal will be reported by the site research team to the CI. Reasons for withdrawal will be anonymously narrated into the study report. Any data collected up until withdrawal will be retained.

Participants who are withdrawn from the study before the 7-day duration will be replaced.

END OF STUDY DEFINITION The end of study is defined as the final data collection for the last recruited participant.

ELIGIBILITY:
Inclusion Criteria

* Children and young people (age 3-15) who are assessed by a Doctor or Dietitian as requiring enteral tube feeding via gastrostomy.
* Children and young people able to receive a minimum of 30% of their daily intake from the study product for at least 7 consecutive days.
* Participant is capable of communication/filling in the questionnaires or having a parent/carer who can answer the questions by close observation of the participant reactions. If there are any communication issues the research dietitian/nurse should support. Written, informed consent from the parent/carer/guardian and assent from the participant obtained.

Exclusion Criteria:

* <3 years old
* >15 years old
* Total Parenteral Nutrition
* Post pyloric enteral feeding
* Enteral tube feeding via Nasogastric tube
* Patients with severe renal, oncology, metabolic, IBD or hepatic conditions who are considered clinically unstable
* Known food allergies or intolerances to any ingredient in the product
* Requirement of a fibre free feed (e.g. IBD)
* Children who had an inability to comply with the study protocol, in the opinion of the investigator
* Children who have been involved in another interventional study within 2 weeks of this study.
* Children with recent changes (within 1 week) in medication used to manage gastrointestinal symptoms

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability with regard to gastrointestinal tolerance | Days 1-7
  Parents/carers will be asked to record gastrointestinal patterns and any symptoms (Diarrhoea, constipation, bloating, nausea, vomiting, burping, flatulence, regurgitation, abdominal pain or discomfort) using a questionnaire.

SECONDARY OUTCOMES:
Ease of use | Day 8
  Parents/carers will be asked to complete a questionnaire using a hedonic scale. (Ease of use is positive if ≥3 )
To test where possible palatability of the Wilbo's Blends+ product. | Day 8
  Palatability is positive (≥5 on the hedonic scale).
Health Care Team perceptions of Wilbo's Blends+. | September 25-March 26
  We will seek feedback from healthcare professionals involved in the study using exploratory qualitative data

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bobo E. Reemergence of Blenderized Tube Feedings: Exploring the Evidence. Nutr Clin Pract. 2016 Dec;31(6):730-735. doi: 10.1177/0884533616669703. Epub 2016 Sep 25. PMID 27646862
- [Background] Marchesi JR, Allen S, Scott E, Jenkins H, Sadlier C, Thomas S. An observational investigation of the faical microbiota and metabonome of gastrostomy fed children, on blended and formula diets. Gut Microbes. 2022 Jan-Dec;14(1):2138661. doi: 10.1080/19490976.2022.2138661. PMID 36284401
- [Background] Shrager S, Adigun A, Motolongo S, Santos CS, Rowe-King P, Duro D. Comparison of Home-Blenderized Formula and Commercial Enteral Formulas for Gastrostomy Tube-Fed Children: A Retrospective, Prospective Cohort Study. Cureus. 2023 Apr 21;15(4):e37944. doi: 10.7759/cureus.37944. eCollection 2023 Apr. PMID 37220453
- [Background] Alabbas F, Dumant C. Outcomes of Blenderized Gastrostomy Feeding in Children at Rouen University Hospital. Pediatric Health Med Ther. 2022 Aug 10;13:271-277. doi: 10.2147/PHMT.S361724. eCollection 2022. PMID 35983160
- [Background] Gallagher K, Flint A, Mouzaki M, Carpenter A, Haliburton B, Bannister L, Norgrove H, Hoffman L, Mack D, Stintzi A, Marcon M. Blenderized Enteral Nutrition Diet Study: Feasibility, Clinical, and Microbiome Outcomes of Providing Blenderized Feeds Through a Gastric Tube in a Medically Complex Pediatric Population. JPEN J Parenter Enteral Nutr. 2018 Aug;42(6):1046-1060. doi: 10.1002/jpen.1049. Epub 2018 Jan 16. PMID 29338077
- [Background] Durnan, S., Kennedy, A., Kennedy, D., Stanley, R., Donohoe, S., Thomas S. & Constable, L. (2021) Practice Toolkit: The Use of Blended Diet with Enteral Feeding Tubes. British Dietetic Association
- [Background] Campbell SM. An anthology of advances in enteral tube feeding formulations. Nutr Clin Pract. 2006 Aug;21(4):411-5. doi: 10.1177/0115426506021004411. PMID 16870811
- [Background] Bonnes SL, Salonen BR, Hurt RT, McMahon MT, Mundi MS. Parenteral and Enteral Nutrition-From Hospital to Home: Will It Be Covered? Nutr Clin Pract. 2017 Dec;32(6):730-738. doi: 10.1177/0884533617734491. Epub 2017 Oct 10. PMID 29016231
- See also: Link to the British Dietetic Association Policy Statement and Practice Toolkit on the use of blended diet with enteral feeding tubes — https://www.bda.uk.com/resource/launch-of-bda-practice-toolkit-the-use-of-blended-diet-with-enteral-feeding-tubes.html
- See also: Home page for Wilbo's Blends — https://wilbosblends.com/